CLINICAL TRIAL: NCT06449794
Title: Neuropsycatric Disorders Among Children With Systemic Lupus Erythematosus in Sohag University Hospital
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amira Mahmoud Ahmed, Resident-pediatric department-sohag hospital university, Sohag University
Other Study IDs: Soh-Med-24-05-10MS
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Anti Phospholipid antibodies — diagnosis of SLE
Radiation: EEG — EEG for Cases with seizures.

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic autoimmune disease involving multiple organs, characterized by the production of autoantibodies and the development of tissue injury. The etiology of SLE is partially known, involving multiple genetic and environmental factors. As many as 50% of patients with SLE have neurological involvement during the course of their disease. Approximately 40% of neuropsychiatric SLE (NPSLE) cases are a consequence of the disease itself; other causes of NPSLE are infections, metabolic disorders, and side effects of drugs. The American College of Rheumatology identified 19 neuropsychiatric syndromes in SLE patients that can be divided into central and peripheral nervous system manifestations. Although this classification includes syndromes with no clear pathophysiological mechanism and is not specific for neuropsychiatric events caused exclusively by SLE, it helps the physician to recognize any neurological involvement . The most common clinical manifestations of juvenile neuropsychiatric SLE (NPSLE) are headache, cognitive dysfunction, mood disturbances and seizures. The pathophysiology of juvenile NPSLE is not yet fully known, but immunological and inflammatory factors, such as autoantibodies, cytokine and prothrombotic states are widely described . The of autoantibodies in the onset of specific clinical manifestations has also been recognized. Juvenile NPSLE manifestations are often difficult to diagnose (. Nineteen neuropsychiatric syndromes have been identified associated with SLE, can be divided into central and peripheral manifestations.

ELIGIBILITY:
Inclusion Criteria:

* The study aims to include all children fulfilling the diagnostic criteria of SLE (The European League Against Rheumatism and The American College of Rheumatology (9)) attending to pediatric rheumatology and immunology clinic at Sohag University Hospitals during the study period.

Exclusion Criteria:

* Children with other rheumatological disorders.; Neonates (infants > 1 month) Children with other neuropsychiatric disorders not attributed to SLE ( e.g. infection, metabolic disorders or side effects of drugs).

Min Age: 1 Year | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study aims to include all children fulfilling the diagnostic criteria of SLE (The European League Against Rheumatism and The American College of Rheumatology (9)) attending to pediatric rheumatology and immunology clinic at Sohag University Hospitals during the study period
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
detect the clinical spectrum of Neuropsycatric disorders in Children with SLE | 1 year
  the diagnostic criteria of SLE (The European League Against Rheumatism and The American College of Rheumatology

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kozora E, Erkan D, West SG, Filley CM, Zhang L, Ramon G, Duggan E, Lockshin MD. Site differences in mild cognitive dysfunction (MCD) among patients with systemic lupus erythematosus (SLE). Lupus. 2013 Jan;22(1):73-80. doi: 10.1177/0961203312468963. PMID 23263866
- [Background] Pamfil C, Fanouriakis A, Damian L, Rinzis M, Sidiropoulos P, Tsivgoulis G, Rednic S, Bertsias G, Boumpas DT. EULAR recommendations for neuropsychiatric systemic lupus erythematosus vs usual care: results from two European centres. Rheumatology (Oxford). 2015 Jul;54(7):1270-8. doi: 10.1093/rheumatology/keu482. Epub 2015 Jan 30. PMID 25638807
- [Background] The American College of Rheumatology nomenclature and case definitions for neuropsychiatric lupus syndromes. Arthritis Rheum. 1999 Apr;42(4):599-608. doi: 10.1002/1529-0131(199904)42:43.0.CO;2-F. PMID 10211873
- [Background] Hanly JG. Diagnosis and management of neuropsychiatric SLE. Nat Rev Rheumatol. 2014 Jun;10(6):338-47. doi: 10.1038/nrrheum.2014.15. Epub 2014 Feb 11. PMID 24514913